CLINICAL TRIAL: NCT01580254
Title: Phase 4 Study to Evaluate Efficacy And Safety of Three Different Preparations of Latanoprost 0,005% Eyedrops in Subjects Affected by Primary Open Angle Glaucoma
Brief Title: Efficacy and Safety of Three Different Latanoprost 0,005% Eyedrops in Subjects Affected by Primary Open Angle Glaucoma
Acronym: LATANOPROST
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Catanzaro (Other)
Responsible Party: Principal Investigator, Luigi Varano, MD - Principal Investigator, M. D., University of Catanzaro
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GENERIC-LATANOPROST
Record Dates: First submitted 2012-04-17; First posted 2012-04-18 (Estimated); Last update posted 2012-04-18 (Estimated); Status verified 2012-04

CONDITIONS: Intraocular Pressure (IOP); Tear Break-Up Time
Keywords: Latanoprost; IOP
MeSH Terms: interventions — Sodium

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- IOPIZE© eyedrops (Active Comparator): subjects will receive a IOP-lowering therapy with latanoprost eyedrops. Drug commercial name is IOPIZE©
  Interventions: Drug: IOPIZE© Latanoprost eyedrops
- GALAXIA© eyedrops (Active Comparator): subjects will receive a IOP-lowering therapy with latanoprost eyedrops. Drug commercial name is GALAXIA©
  Interventions: Drug: GALAXIA© Latanoprost eyedrops
- Latanoprost RATIOPHARM© eyedrops (Active Comparator): subjects will receive a IOP-lowering therapy with latanoprost eyedrops. Drug commercial name is Latanoprost RATIOPHARM©
  Interventions: Drug: Latanoprost RATIOPHARM© latanoprost eyedrops

INTERVENTIONS:
Drug: IOPIZE© Latanoprost eyedrops — patients will receive in each eligible eye one drop of IOPIZE© Latanoprost eyedrops once a day, in the evening (8pm), for two months
  Other Names: IOPIZE© eyedrops (S.I.F.I. S.p.A. - Aci S. Antonio (CT), Italy); authorization numbers:; 039276011; 039276023; 039276035
  Arms: IOPIZE© eyedrops
Drug: GALAXIA© Latanoprost eyedrops — patients will receive in each eligible eye one drop of GALAXIA© Latanoprost eyedrops once a day, in the evening (8pm), for two months
  Other Names: GALAXIA© eyedrops (ALFA INTES Industria Terapeutica Splendore S.r.l. - Casoria (NA), Italy); authorization number:; 038622015
  Arms: GALAXIA© eyedrops
Drug: Latanoprost RATIOPHARM© latanoprost eyedrops — patients will receive in each eligible eye one drop of Latanoprost RATIOPHARM© Latanoprost eyedrops once a day, in the evening (8pm), for two months
  Other Names: Latanoprost RATIOPHARM© eyedrops (RATIOPHARM GmbH - Ulm, Germany); authorization number:; 039468018/M
  Arms: Latanoprost RATIOPHARM© eyedrops

SUMMARY:
This study examines efficacy and tolerability of 3 different Latanoprost 0.005% eyedrops preparations, commercially available in Italy, in subjects affected by primary open angle glaucoma.

DETAILED DESCRIPTION:
Prospective, randomized, single blinded study of the duration of 3 months, involving subjects affected by POAG or OH under therapy with different Latanoprost drugs (Galaxia, Iopize or Latanoprost Rathiopharm).

A total of 120 patients affected by POAG or OH newly diagnosed or already under topical therapy. will be recruited.

After a recruitment visit to assest eligibility of each subject, a "run-in" therapy composed of timolol 0,5% 2 drops per day will be prescribed for 4 weeks.

Then a baseline visit will be performed to evaluate IOP values and adverse effects in each subject. All subjects elegible for a therapy with a single dose of Latanoprost will be randomized into 3 arms.

After 4 weeks of therapy a second visit will be made to assest IOP changes and safety. Therapy will be continued for another 4 weeks, and after that, a final visit will be made.

ELIGIBILITY:
Inclusion Criteria:

* Age ranged between 18 and 80
* Untreated IOP ranged between 21 and 30 mmHg
* IOP already treated with a single drug (monotherapy) ranged between 10 and 28 mmHg

Exclusion Criteria:

* History of adverse events or any controindication to drugs administred during sperimentation, i. e. Latanoprost and Timolol.
* Narrow or closed iridocorneal angle.
* History of acute angle-closure glaucoma.
* Previous laser trabeculoplasty within 3 months before screening.
* Severe visual field defects within 10° from fixation in at least one eye (at least 2 points with a p<0,5 in a pattern deviation map obtained from a reliable 24-2 Sita Standard SAP).
* History of refractive surgery or any keratoplasty procedure, corneal opacities or diseases that make not suitable applanation tonometry.
* Use of contact lenses.
* BCVA less than 20/200.
* Ocular inflammation/infection occurring within three months before screening.
* History of bradicardia, systemic hypotension, bundle branch or any atrio-ventricular block
* Asthma
* Women of childbearing potential who were not using adequate contraceptive methods or who were pregnant or nursing

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2011-06; Primary Completion 2012-06 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
intraocular pressure (IOP) in mmHg | one month - two months
  to evaluate intraocular pressure (IOP) reduction after one and two months treatment with latanoprost eyedrops

SECONDARY OUTCOMES:
Tear Break-Up Time (BUT) expressed in seconds | one month - two months
  After one and two months of therapy with latanoprost, tear BUT will be calculated, through the use of fluoresceine staining of the tear film.

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Varano, M. D., Principal Investigator — University of Catanzaro
Locations (1):
- University of Catanzaro - Eye Department, Catanzaro, Catanzaro, Italy